CLINICAL TRIAL: NCT02868710
Title: The Incidence of Training Responsiveness to Cardiorespiratory Fitness and Cardiometabolic Measurements Following Individualized and Standardized Exercise Prescription
Brief Title: Individual Variability to Aerobic Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Colorado University (Other)
Responsible Party: Principal Investigator, Lance Dalleck, Associate Professor, Western Colorado University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WeternStateCU
Record Dates: First submitted 2016-08-09; First posted 2016-08-16 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Cardiovascular Disease
Keywords: primary prevention
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Individualized method (Experimental): 3 days a week of exercise at the following intensity and energy expenditure:
  Week 1: HR > VT1; 5.6 kcal/kg/wk Week 2: HR > VT1; 8.4 kcal/kg/wk Week 3: HR > VT1; 11.2 kcal/kg/wk Week 4: HR ≥ VT1 to <VT2; 11.2 kcal/kg/wk Week 5-6: HR ≥ VT1 to <VT2; 11.2 kcal/kg/wk Week 7: HR ≥ VT1 to <VT2; 12.6 kcal/kg/wk Week 8: HR ≥ VT1 to <VT2; 14 kcal/kg/wk Week 9-10: HR ≥ VT2; 14 kcal/kg/wk Week 11-12: HR ≥ VT2; 15.4 kcal/kg/wk
  Interventions: Other: Exercise
- Standardized method (Experimental): 3 days a week of exercise at the following intensity and energy expenditure:
  Week 1: 40-45% HRR; 5.6 kcal/kg/wk Week 2: 40-45% HRR; 8.4 kcal/kg/wk Week 3: 40-45% HRR; 11.2 kcal/kg/wk Week 4: 50-55% HRR; 11.2 kcal/kg/wk Week 5-6: 55-60% HRR; 11.2 kcal/kg/wk Week 7: 55-60% HRR; 12.6 kcal/kg/wk Week 8: 55-60% HRR; 14 kcal/kg/wk Week 9-10: 60-65% HRR; 14 kcal/kg/wk Week 11-12: 60-65% HRR; 15.4 kcal/kg/wk
  Interventions: Other: Exercise
- Control (No Intervention): non-exercise control group
  Testing at baseline and post-program (12 weeks)

INTERVENTIONS:
Other: Exercise — Continuous aerobic exercise prescribed according to two exercise intensity methods: individualized (i.e. ventilatory threshold) and standardized (i.e. heart rate reserve)
  Arms: Individualized method; Standardized method

SUMMARY:
The purpose of this study is to: 1) determine the cohort specific technical error to use in the categorization of response rate; 2) determine if an individualized intensity prescription is superior to a standard approach in regards to VO2max and cardiometabolic risk factor responsiveness; 3) Investigate the time course changes throughout 12 weeks of CRF training between an individualized and standardized exercise prescription; and 4) determine if non-responders can become responders if the exercise intensity prescription is modified.

It is hypothesized that:

1. The individualized method will elicit a greater responsiveness for all measurements when compared to the standardized method.
2. There will be a greater amount of non-responders in the standardized group (based on changes in VO2max).
3. When participants in the standardized group are considered non-responders and change their exercise prescription to the individualized group, they will become a responder (based on changes in VO2max)

DETAILED DESCRIPTION:
It has generally been accepted there is individual variability to cardiorespiratory fitness (CRF) training. However, the underlying cause of the variability is not well understood. Traditionally, a standardized approach to exercise prescription has utilized relative percentages of maximal heart rate (HR), HR reserve (HRR), maximal oxygen consumption (VO2max), or VO2 reserve to establish exercise intensity. This 'one size fits all' model fails to take into consideration individual metabolic responses to exercise and may be related to the variability in training responses.

An individualized exercise prescription utilizing a threshold-based training model (i.e. ventilatory threshold) would help consider individual metabolic responses to exercise training. However, minimal research has been conducted to differentiate between the standardized and individualized methods. Therefore, a randomized control trial within a community-based wellness program will be implemented to investigate the following research question: does an individualized exercise prescription decrease the incidence of non-response to CRF and cardiometabolic measurements compared to the standardized approach? The criteria to determine the incidence of response will be set based on the biological variability and measurement error determined during baseline testing.

A secondary outcome of the study will be investigating the time course changes in response to 12 weeks of individualized and standardized exercise prescription. Currently, minimal research exists on the effects of differing exercise prescription and the time course changes with the reporting of individual data.

Many experimental trials are conducted in a very controlled and supervised environment and may lack real world application. This investigation would occur in a community-based wellness program to encourage a 'real-world' application. Results of this study would enhance the ability of exercise physiologists to prescribe exercise to the individual, rather than a 'one size fits all' model. This would be the first study to investigate individualized versus standardized exercise prescription with an isocaloric exercise volume.

Therefore, sedentary men and women (n = 40) will be randomized to one of two experimental groups - individualized or standardized. There will be a separate control group (n = 20) that is recruited from the community that has the same inclusion criteria as the experimental group. Exercise training will be performed 3 days a week with weekly energy expenditure progressively increasing from 5.6 to 15.4 kcal/kg/week for 12 weeks with one of two exercise intensity regimens: 1) a standardized method based on percentages of HRR, or 2) a threshold based method with the use of the first (VT1) and second ventilatory threshold (VT2). Participants will undergo testing (anthropometric measures, blood profile, and maximal exercise test) at baseline, 4 weeks, 8 weeks, and 12 weeks.

Following the 12 week intervention, participants will be categorized as a responder or non-responder based on overall changes in VO2max. For responders, they will be done with the intervention. However, non-responders will be asked to complete a second 12 week intervention in the other experimental group (i.e. a non-responder in the standardized group will now complete a 12 week intervention the individualized group. The exercise prescription and progression will be the same for the second 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Considered low to moderate risk for cardiovascular disease based on the American College of Sports medicine guidelines
* Currently sedentary (participating in less than 30 minutes of moderate intensity physical activity on at least three days a week)
* Resided at an altitude of 2300 meters for at least the last 6 months

Exclusion Criteria:

* Any known sign, symptom, or diagnosed cardiovascular, pulmonary, metabolic, or similar disease

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-09; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Maximal Oxygen Uptake (VO2max) | 12 weeks

SECONDARY OUTCOMES:
Total cholesterol | 12 weeks
Low-density lipoprotein | 12 weeks
High-density lipoprotein | 12 weeks
Triglycerides | 12 weeks
Fasting blood glucose | 12 weeks
Waist circumference | 12 weeks
Height | 12 weeks
Weight | 12 weeks
Resting heart rate | 12 weeks
Resting blood pressure | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Western State Colorado University, Gunnison, Colorado, United States

REFERENCES:
- [Derived] Weatherwax RM, Harris NK, Kilding AE, Dalleck LC. The incidence of training responsiveness to cardiorespiratory fitness and cardiometabolic measurements following individualized and standardized exercise prescription: study protocol for a randomized controlled trial. Trials. 2016 Dec 19;17(1):601. doi: 10.1186/s13063-016-1735-0. PMID 27993169